CLINICAL TRIAL: NCT01396525
Title: A Prospective, Non-randomized, Two Arm, Multi-center Clinical Trial to Evaluate the Safety and Efficacy of the Absolute Pro™ Peripheral Self-Expanding Stent System and the Omnilink Elite™ Peripheral Balloon-Expandable Stent System in Subjects With Atherosclerotic de Novo or Restenotic Lesions in the Native Common Iliac Artery and/or Native External Iliac Artery.
Brief Title: Trial to Evaluate the Safety & Efficacy of the Omnilink Elite™ Peripheral Balloon-Expandable Stent System in Subjects With Atherosclerotic de Novo or Restenotic Lesions in the Native Common Iliac Artery and/or Native External Iliac Artery
Acronym: MOBILITY OE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-107 Omnilink Elite Arm (OE); 08-107 AP, NCT00844532 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Vascular Disease
Keywords: Atherosclerosis; Peripheral artery disease; Peripheral vascular disease; PAD; Claudication; Peripheral Arterial Occlusive Disease; Stent; PAOD; PVD
MeSH Terms: conditions — Peripheral Vascular Diseases; Atherosclerosis; Peripheral Arterial Disease; Intermittent Claudication; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omnilink Elite™ Peripheral Balloon-Expandable Stent System (Experimental)
  Interventions: Device: Omnilink Elite™ Peripheral Balloon-Expandable Stent System

INTERVENTIONS:
Device: Omnilink Elite™ Peripheral Balloon-Expandable Stent System — Patients with treatment of a maximum of two bilateral de novo or restenotic atherosclerotic lesions in the native common iliac artery and/or native external iliac artery (one lesion per side).

SUMMARY:
To determine the safety and efficacy of the Omnilink Elite™ Peripheral Balloon-Expandable Stent System in subjects with atherosclerotic de novo or restenotic lesions in the native common iliac artery and/or native external iliac artery.

DETAILED DESCRIPTION:
The MOBILITY study was a prospective, non-randomized, two-arm, multi-center study. The 2 arms (Omnilink Elite arm and Absolute Pro arm) were designed to independently assess the safety and effectiveness of the 2 devices used in this study.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject must be at least 18 and < 90 years of age.
2. Subject has been informed of the nature of the trial, agrees to its provisions, and has signed the informed consent form.
3. Subject must agree to undergo all protocol-required follow-up examinations and requirements at the investigational site.
4. History of symptomatic claudication (Rutherford Becker Clinical Category 2-3) or ischemic rest pain (Rutherford Becker Clinical Category 4).
5. Female subjects of childbearing potential must have had a negative pregnancy test before treatment, and must not be nursing at the time of treatment, and agree at time of consent to use birth control during participation in this trial up to and including the follow-up at 9 months.

Angiographic Inclusion Criteria

1. Up to two bilateral de novo or restenotic lesions of the native common iliac artery and/or native external iliac artery may be treated(one per side).
2. Common iliac artery lesion visually estimated to be ≥50% stenosis and ≤100% stenosis (total occlusion)
3. External iliac artery lesion visually estimated to be ≥50% stenosis and ≤99% stenosis
4. Lesion length for stenosis of the common or external iliac artery visually estimated to be ≥ 10 mm and ≤ 110 mm (Absolute Pro)
5. Lesion length for total occlusion of the common iliac artery visually estimated to be ≤40 mm
6. Target vessel reference diameter visually estimated to be ≥3.6 mm and ≤9.1 mm (Absolute Pro)
7. On the treatment side(s), patent superficial femoral and popliteal arteries and at least one patent distal outflow artery with in-line distal vessel flow to the foot as confirmed by arteriography. Patent is defined as < 50% stenosis.
8. Lesion length for stenosis of the common or external iliac artery visually estimated to be ≥ 10 mm and ≤ 50 mm (Omnilink Elite).
9. Target vessel reference diameter visually estimated to be ≥ 5.0 mm and ≤ 11.0 mm (Omnilink Elite).

Clinical Exclusion Criteria

1. Subject is unable to walk.
2. Subject has had recent major surgery (last 3 months) e.g., abdominal surgery, coronary artery bypass graft surgery, thoracic surgery.
3. Subject has received, or is on the waiting list for a major organ transplant (heart, lung, kidney, liver).
4. Subject is diagnosed as Rutherford Becker Clinical Category 0, 1, 5, or 6.
5. Subject has ulcers or lesions on the lower extremity(ies) of the target lesion side(s).
6. Subject has elevated serum creatinine > 2.0 mg/dl.
7. Subject has uncontrolled diabetes mellitus (DM) (serum glucose > 400 mg/dl).
8. Subject has had a myocardial infarction(MI)(Q-wave or NQWMI) within the previous 30 days.
9. Subject has had a stroke within the previous 30 days and/or has deficits from a prior stroke that limits the subjects ability to walk.
10. Subject has unstable angina defined as rest angina with ECG changes.
11. Subject has a groin infection, or an acute systemic infection that is currently under treatment.
12. Subject has acute thrombophlebitis or deep vein thrombosis in either extremity.
13. Subject requires any planned procedure within 30 days after the index procedure that would necessitate the discontinuation of aspirin, clopidogrel or ticlopidine following the procedure.
14. Subject has other medical illnesses (e.g., cancer or congestive heart failure) that may cause the subject to be non-compliant with protocol requirements, confound the data interpretation, or is associated with limited life-expectancy (i.e., less than 2 years).
15. Subject is currently participating in an investigational drug or device trial that has not completed the primary endpoint follow-up or that clinically interferes with the current trial endpoints.
16. Subject is unable to understand or unwilling to cooperate with trial procedures or is unwilling or unable to return to the treatment center for follow-up visits.
17. If intended stent is Absolute Pro, subject has known hypersensitivity or contraindication to nickel, titanium or platinum; subject has known hypersensitivity or contraindication to standard intraprocedure anticoagulant(s); subject has sensitivity to contrast which cannot be adequately pre-treated with medication.
18. Subject has known allergy or contraindication to aspirin or clopidogrel (Plavix®); if allergy or contraindication is to clopidogrel, subject is unable to tolerate ticlopidine (Ticlid®).
19. Subject has known bleeding disorder or hypercoagulable disorder, or will refuse blood transfusions.
20. Subject has suffered a gastrointestinal (GI) bleed within 30 days before the index procedure that would interfere with antiplatelet therapy.
21. If intended stent is Omnilink Elite, subject has known hypersensitivity or contraindication to cobalt chromium; subject has known hypersensitivity or contraindication to standard intraprocedure anticoagulant(s); subject has sensitivity to contrast which cannot be adequately pre-treated with medication.
22. Requirement of general anesthesia or spinal block for the procedure.
23. Presence of contralateral limb amputation that was performed to treat any non-traumatic disease in that limb, e.g. atherosclerotic, vascular, neuropathic.
24. Presence of bypass conduit in any outflow vessel, i.e. SFA, popliteal, anterior tibial, posterior tibial, peroneal, ipsilateral to the target lesion.
25. Subject requires a concomitant percutaneous endovascular procedure in another vessel, e.g. coronary.
26. Target lesion is in an iliac artery that has been previously stented.

Angiographic Exclusion Criteria

1. Subject has a totally occluded (100% stenosis) external iliac artery ipsilateral to the target lesion.
2. Subject has a totally occluded (100% stenosis) outflow artery (SFA) ipsilateral to the target lesion
3. Target lesion is within or adjacent to an aneurysm.
4. Lesion is located within or beyond a vessel that contains a bypass graft.
5. Lesion(s) requires atherectomy (or ablative devices) to facilitate stent delivery.
6. Subject has a history of aortic revascularization or has an abdominal aortic aneurysm > 3cm.
7. Lesion extends beyond the inguinal ligament.
8. Subject has angiographic evidence of thrombus in the target disease segment or vessel that is unresponsive to anti-thrombotic therapies.
9. Subject has multilevel disease in the target extremity that requires other staged procedures within 30 days before or after the procedure.
10. On the treatment side(s), subject is without patent superficial femoral and popliteal arteries and at least one patent distal outflow artery with in-line distal vessel flow to the foot as confirmed by arteriography. Patent is defined as < 50% stenosis.
11. Requirement for > 1 stent to treat full length of lesion.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony S. Das, MD, Principal Investigator — Presbyterian Heart Institute, Dallas, TX; Manish Mehta, MD, MPH, Principal Investigator — Albany Medical Center, Albany, NY.
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with chronic lower extremity peripheral arterial disease (PAD) admitted for percutaneous CIA or EIA revascularization were screened for eligibility. Subjects who met all general and clinical eligibility criteria, and signed the informed consent, underwent arteriography of the target iliac artery.
Groups:
- Omnilink Elite™ Peripheral Balloon-Expandable Stent System: Omnilink Elite™ Peripheral Balloon-Expandable Stent System : Patients with treatment of a maximum of two bilateral de novo or restenotic atherosclerotic lesions in the native common iliac artery and/or native external iliac artery (one lesion per side).
Period: Overall Study
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Started | 153
Completed | 127
Not Completed | 26
Not completed — Withdrawal by Subject | 8
Not completed — Death | 14
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 88
Region of Enrollment [Number; unit: participants]
  United States | 153

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event (MAE)
Description: Defined as death, myocardial infarction (MI), clinically-driven target lesion revascularization, and limb loss (major amputation only) on the treated side(s).
Time Frame: 9 months
Population: Intent to treat (ITT) population. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 149
percentage of participants | 5.4 [NA to 9.5] — One-sided 95% confidence interval was computed for this endpoint, lower bound is not provided.

2. Secondary Outcome: Device Success
Description: On a per device basis, the achievement of successful delivery and deployment of the trial device(s) at the intended location(s) and successful withdrawal of the delivery catheter(s).
Time Frame: Acute: from beginning of index procedure to end of procedure
Population: ITT population, per device analysis. Included 210 stents plus 1 stent inserted but not implanted due to device malfunction, 2 stents excluded due to inappropriate sizing (stents were not implanted), 1 stent excluded as stent was not implanted per physician's choice and had no device malfunction.
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: devices
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (devices) | 211
percentage of devices | 98.6 [95.9 to 99.7]

3. Secondary Outcome: Technical Success
Description: Technical success is defined as device success (the achievement of successful delivery and deployment of the trial device(s) at the intended target lesion(s), successful withdrawal of the delivery catheter(s)), and attainment of a final residual stenosis of < 30% by QA or as reported by the investigator.
Time Frame: Acute: from beginning of index procedure to end of procedure
Population: ITT population, per lesion analysis
Measure: Number (95% Confidence Interval); unit: percentage of target lesions
Units Other Than Participants: target lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (target lesions) | 203
percentage of target lesions | 93.1 [88.7 to 96.2]

4. Secondary Outcome: Procedure Success
Description: Procedure success is defined as technical success (device success and attainment of a final residual stenosis of < 30% by QA) without complications within two (2) days after the index procedure or at hospital discharge, whichever is sooner.
Time Frame: Beginning of index procedure to 2 days post-index procedure or discharge, whichever is sooner
Population: ITT population, per subject analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 91.5 [85.9 to 95.4]

5. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: The thigh brachial index is the ratio of the resting ipsilateral thigh systolic blood pressure as compared to the highest resting brachial systolic blood pressure. A normal range is 0.9 to 1.3.
Time Frame: Pre-procedure
Population: ITT population, per limb analysis. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 141
Number analyzed (Limbs) | 189
Ratio | 0.9 (0.2)

6. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: Post-Procedure
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 141
Number analyzed (Limbs) | 188
Ratio | 1.0 (0.2)

7. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 1 month
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 133
Number analyzed (Limbs) | 178
Ratio | 1.0 (0.1)

8. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 9 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 136
Number analyzed (Limbs) | 180
Ratio | 1.0 (0.2)

9. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 2 years
Population: ITT population, per limb analysis.The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 106
Number analyzed (Limbs) | 140
Ratio | 1.0 (0.1)

10. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 3 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 96
Number analyzed (Limbs) | 132
Ratio | 1.0 (0.2)

11. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: The changes in thigh brachial index is the absolute change between the pre-procedure measure and the stated timepoint measure.
Time Frame: Between baseline and Post-procedure
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 133
Number analyzed (Limbs) | 179
Ratio | 0.2 (0.2)

12. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 11
Time Frame: Between Baseline and 1 month
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 125
Number analyzed (Limbs) | 168
Ratio | 0.2 (0.2)

13. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 11
Time Frame: Between baseline and 9 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 124
Number analyzed (Limbs) | 166
Ratio | 0.1 (0.2)

14. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: The changes in thigh brachial index is the ratio of change between the pre-procedure measure and the stated timepoint measure.
Time Frame: Between baseline and 2 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 96
Number analyzed (Limbs) | 128
Ratio | 0.2 (0.2)

15. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 14
Time Frame: Between baseline and 3 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 87
Number analyzed (Limbs) | 122
Ratio | 0.2 (0.2)

16. Secondary Outcome: Walking Impairment Questionaire Scores
Description: Measured by the Walking Impairment Questionnaire (WIQ), a disease-specific instrument utilized to characterize walking ability through a questionnaire as an alternative to treadmill testing. It is a measure of subject-perceived walking performance for subjects with Peripheral Artery Disease (PAD) and/or intermittent claudication. The WIQ quantifies patient-reported walking speed, walking distance, and stair-climbing ability, respectively, on a scale of 0 (= worst) to 100 (= best). The highest possible score for each domain is 100%, which indicates no difficulty. Lowest possible score for each domain is 0%, which indicates inability to perform the activity.
Time Frame: Pre-procedure
Population: ITT population, per subject analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Walking Distance Score; Walking Speed Score; Stair Climbing Score: Omnilink Elite™ Peripheral Balloon-Expandable Stent System : Patients with treatment of a maximum of two bilateral de novo or restenotic atherosclerotic lesions in the native common iliac artery and/or native external iliac artery (one lesion per side).
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 152 | 151 | 151
score on a scale | 17.5 (22.7) [17.5 to 22.7] | 20.1 (24.0) | 26.0 (25.8)

17. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 16
Time Frame: 1 month
Population: ITT population, per subject analysis. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 131 | 131 | 129
score on a scale | 56.4 (38.0) | 50.4 (34.4) | 56.1 (36.7)

18. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 16
Time Frame: 9 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 138 | 138 | 134
score on a scale | 56.6 (38.6) | 47.6 (33.2) | 60.4 (35.9)

19. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 16
Time Frame: 2 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 112 | 113 | 112
score on a scale | 49.1 (37.9) | 44.5 (31.1) | 51.7 (33.8)

20. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 16
Time Frame: 3 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 107 | 107 | 105
score on a scale | 46.8 (37.1) | 41.8 (30.4) | 55.4 (34.9)

21. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: The Rutherford Becker clinical category is a scale to measure chronic limb ischemia.
  Category and Clinical Description:
  0 = Asymptomatic, no hemodynamically significant occlusive disease, 1 = Mild claudication, 2 = Moderate claudication, 3 = Severe claudication, 4 = Ischemic rest pain, 5 = tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, 6 = Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable
Time Frame: Pre-Procedure
Population: as for outcome 5
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limb(s)
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limb(s)) | 203
percentage of target limbs
  0 | 0.0
  1 | 0.0
  2 | 43.8
  3 | 54.7
  4 | 1.5
  5 | 0.0
  6 | 0.0

22. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 1 month
Population: as for outcome 9
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 134
Number analyzed (limbs) | 180
percentage of target limbs
  0 | 57.8
  1 | 23.9
  2 | 15.0
  3 | 3.3
  4 | 0.0
  5 | 0.0
  6 | 0.0

23. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 9 months
Population: as for outcome 5
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 137
Number analyzed (limbs) | 182
percentage of target limbs
  0 | 59.9
  1 | 23.6
  2 | 11.5
  3 | 4.4
  4 | 0.5
  5 | 0.0
  6 | 0.0

24. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 2 years
Population: as for outcome 5
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 108
Number analyzed (limbs) | 143
percentage of target limbs
  0 | 66.0
  1 | 16.0
  2 | 15.3
  3 | 2.8
  4 | 0.0
  5 | 0.0
  6 | 0.0

25. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 3 years
Population: as for outcome 5
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 101
Number analyzed (limbs) | 138
percentage of target limbs
  0 | 64.0
  1 | 16.5
  2 | 15.1
  3 | 3.6
  4 | 0.0
  5 | 0.0
  6 | 0.7

26. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: Change in Rutherford Becker Clinical Category:
  Worsening Rutherford Becker Clinical Category:
  Deterioration (an increase) in the Rutherford Becker Clinical Category by at least two categories from baseline and subsequently from the earliest post-procedural measurement or to a category 5 or 6.
  Improved Rutherford Becker Clinical Category:
  An improvement (a decrease) in the Rutherford Becker Clinical Category of at least one category from baseline and subsequently from the earliest post-procedural measurement.
Time Frame: Between baseline and 1 month
Population: as for outcome 5
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 134
Number analyzed (Limbs) | 180
percentage of target limbs
  Improved by >/= 3 categories | 36.1
  Improved by 2 categories | 34.4
  Improved by 1 category | 18.9
  No change | 8.9
  Worsened by 1 category | 1.7
  Worsened by 2 categories | 0.0
  Worsened by 3 categories or more | 0.0

27. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 26
Time Frame: Between baseline and 9 months
Population: as for outcome 5
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 137
Number analyzed (Limbs) | 182
percentage of target limbs
  Improved by >/= 3 categories | 34.6
  Improved by 2 categories | 41.2
  Improved by 1 category | 13.2
  No change | 7.1
  Worsened by 1 category | 3.8
  Worsened by 2 categories | 0.0
  Worsened by 3 categories or more | 0.0

28. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 26
Time Frame: Baseline and 2 years
Population: as for outcome 9
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 108
Number analyzed (Limbs) | 143
percentage of target limbs
  Improved by >/= 3 categories | 35.4
  Improved by 2 categories | 37.5
  Improved by 1 category | 16.7
  No change | 9.0
  Worsened by 1 category | 1.4
  Worsened by 2 categories | 0.0
  Worsened by >/= 3 categories | 0.0

29. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 26
Time Frame: Baseline and 3 years
Population: as for outcome 9
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 101
Number analyzed (Limbs) | 138
percentage of target limbs
  Improved by >/= 3 categories | 38.8
  Improved by 2 categories | 33.1
  Improved by 1 category | 15.1
  No Change | 11.5
  Worsened by 1 category | 0.7
  Worsened by 2 categories | 0.0
  Worsened by >/= 3 categories | 0.7

30. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years.Target lesion revascularization (TLR) is defined as any revascularization at the target lesion with or without evidence of target lesion diameter stenosis ≥ 50% determined by Duplex ultrasonography (DUS) or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion).
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions
  1 month | 99.0
  9 months | 95.5

31. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. Target lesion revascularization (TLR) is defined as any revascularization at the target lesion with or without evidence of target lesion diameter stenosis ≥ 50% determined by DUS or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion).
Time Frame: 18 months
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this time point.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions | 93.9

32. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: as for outcome 31
Time Frame: 2 years
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this time point.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions | 90.5

33. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: as for outcome 31
Time Frame: 3 years
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this time point.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions | 87.6

34. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years. Clinically-driven is defined as: Revascularization of the stent with evidence of new distal ischemic signs (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion, and target lesion diameter stenosis ≥ 50% determined by duplex ultrasound or arteriography.) (Note: This does not include coincidental overlap of a percutaneous transluminal angioplasty (PTA) balloon or stent into a study stent, that has <50% stenosis, while treating a non-target lesion in the target vessel).
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions
  1 month | 99.5
  9 months | 97

35. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. Clinically-driven TLR is defined as: Revascularization of the stent with evidence of new distal ischemic signs (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion, and target lesion diameter stenosis ≥ 50% determined by duplex ultrasound or arteriography.) (Note: This does not include coincidental overlap of a PTA balloon or stent into a study stent, that has <50% stenosis, while treating a non-target lesion in the target vessel).
Time Frame: 18 months
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this time point.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions | 95.3

36. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: as for outcome 35
Time Frame: 2 years
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this time point.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions | 93.1

37. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: as for outcome 35
Time Frame: 3 years
Population: ITT population. This analysis represents those subjects with target lesions who were event free at this time point.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target lesions | 90.8

38. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. Target Vessel Revascularization (TVR) is defined as any revascularization of the target vessel, outside of the target lesion, with or without evidence of diameter stenosis ≥ 50% determined by DUS or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target vessel).
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects with lesions in target vessels who were event free at this timepoint
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (lesions) | 203
percentage of target vessels
  1 month | 99.0
  9 months | 98.5

39. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 38
Time Frame: 18 months
Population: ITT population. This analysis represents those subjects with lesions in target vessels who were event free at this time point.
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target vessels | 98.0

40. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 38
Time Frame: 2 years
Population: as for outcome 39
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target vessels | 97.4

41. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 38
Time Frame: 3 years
Population: as for outcome 39
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target vessels | 95.6

42. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Vessel Revascularization (CD-TVR) for the Treated Limb(s)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. Clinically-driven Target Vessel Revascularization is defined as revascularization of the target vessel (outside the target lesion) with evidence of new distal ischemic signs (worsening Rutherford Becker clinical category that is clearly referable to the target vessel, and diameter stenosis ≥ 50% determined by DUS or arteriography).
Time Frame: 1 month and 9 months
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (lesions) | 203
percentage of target vessels
  1 month | 99.5
  9 months | 99.5

43. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 42
Time Frame: 18 months
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target vessels | 99

44. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically Driven Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 42
Time Frame: 2 years
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target vessels | 98.4

45. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically DrivenTarget Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 42
Time Frame: 3 years
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (Lesions) | 203
percentage of target vessels | 96.6

46. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. Target extremity revascularization (TER) is defined as any revascularization of a target extremity vessel (distal to the superior border of the inguinal ligament on the ipsilateral side) with or without evidence of vessel diameter stenosis ≥ 50% determined by DUS or arteriography, and with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category).
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects with vessels in the extremity with the target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of limbs
  1 month | 99.5
  9 months | 98.0

47. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: as for outcome 46
Time Frame: 18 months
Population: as for outcome 46
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of limbs | 95.8

48. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: as for outcome 46
Time Frame: 2 years
Population: as for outcome 46
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of limbs | 94.1

49. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: as for outcome 46
Time Frame: 3 years
Population: as for outcome 46
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of limbs | 94.1

50. Secondary Outcome: Primary Stent Patency
Description: Absence of in-stent restenosis of the target lesion (≥50%) as determined by duplex ultrasound or angiogram and without interval reintervention since the initial study procedure.
Time Frame: 1 month
Population: ITT population, per lesion analysis. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 141
Number analyzed (limbs) | 188
percentage of limbs | 97.3

51. Secondary Outcome: Primary Stent Patency
Description: as for outcome 50
Time Frame: 9 months
Population: as for outcome 50
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 137
Number analyzed (limbs) | 179
percentage of limbs | 89.9

52. Secondary Outcome: Primary Stent Patency
Description: as for outcome 50
Time Frame: 2 years
Population: as for outcome 50
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 123
Number analyzed (limbs) | 163
percentage of limbs | 76.7

53. Secondary Outcome: Primary Stent Patency
Description: as for outcome 50
Time Frame: 3 years
Population: as for outcome 50
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 118
Number analyzed (Limbs) | 155
percentage of limbs | 68.4

54. Secondary Outcome: Restenosis
Description: Defined as ≥ 50% stenosis at follow-up.
Time Frame: 9 months
Population: ITT population. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Number (95% Confidence Interval); unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 137
Number analyzed (limbs) | 185
percentage of limbs | 9.7 [5.9 to 14.9]

55. Secondary Outcome: Restenosis
Description: Defined as ≥ 50% stenosis at follow-up.
Time Frame: 2 years
Population: as for outcome 54
Measure: Number (95% Confidence Interval); unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 121
Number analyzed (limbs) | 159
percentage of limbs | 20.8 [14.7 to 27.9]

56. Secondary Outcome: Restenosis
Description: Defined as ≥ 50% stenosis at follow-up.
Time Frame: 3 years
Population: as for outcome 54
Measure: Number (95% Confidence Interval); unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 113
Number analyzed (limbs) | 148
percentage of limbs | 27.0 [20.1 to 34.9]

57. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects who were event free at this timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants
  1 month | 100
  9 months | 99.3

58. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years.
Time Frame: 18 months
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 94.5

59. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years.
Time Frame: 2 years
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 93.8

60. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years.
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 90.2

61. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. The term myocardial infarction should be used when there is evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia.
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects who were event free at this timepoint
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants
  1 month | 100.0
  9 months | 99.3

62. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: as for outcome 61
Time Frame: 18 months
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 97.2

63. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: as for outcome 61
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 95.7

64. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: as for outcome 61
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 95.7

65. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years. The removal of a body extremity by surgery. For this study, the definition of amputation will only include amputations of the limb(s) that was/were treated. A major amputation will be defined as at or above the ankle.
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this timepoint
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs
  1 month | 100.0
  9 months | 100.0

66. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. The removal of a body extremity by surgery. For this study, the definition of amputation will only include amputations of the limb(s) that was/were treated. A major amputation will be defined as at or above the ankle.
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs | 100

67. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: as for outcome 66
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs | 100

68. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: as for outcome 66
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs | 99.4

69. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. Embolism is the formation of a thrombus within the target lesion or stent with migration or atherosclerotic emboli migration to a distal artery.
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects who were event free at this timepoint
Measure: Number; unit: percentage of particpants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of particpants
  1 month | 99.3
  9 months | 98.0

70. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: as for outcome 69
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects who were event free at this timepoint
Measure: Number; unit: percentage of particpants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of particpants | 98

71. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: Outcome measure analyzed at 1 and 9 months and at 2 and 3 years. Embolism is the formation of a thrombus within the target lesion or stent with migration or atherosclerotic emboli migration to a distal artery.
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 97.3

72. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: as for outcome 71
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
percentage of participants | 96.5

73. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Minor) of the Treated Limb(s)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years. The removal of a body extremity by surgery. For this study, the definition of amputation will only include amputations of the limb(s) that was/were treated. A minor amputation will be defined as below the ankle.
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this timepoint
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs
  1 month | 100.0
  9 months | 100.0

74. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Minor) of the Treated Limb(s)
Description: Outcome measure analyzed at 1, 9 and 18 months, 2 and 3 years. The removal of a body extremity by surgery. For this study, the definition of amputation will only include amputations of the limb(s) that was/were treated. A minor amputation will be defined as below the ankle.
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs | 100.0

75. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Minor) of the Treated Limb(s)
Description: as for outcome 74
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs | 100.0

76. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Minor) of the Treated Limb(s)
Description: as for outcome 74
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of target limbs
Units Other Than Participants: limbs
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 153
Number analyzed (limbs) | 203
percentage of target limbs | 99.4

77. Secondary Outcome: Stent Thrombosis
Description: Defined as a total occlusion documented by duplex ultrasound and/or arteriography at the stent site with or without symptoms that occurs ≤ 30 days post index procedure.
Time Frame: 1 month
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: percentage of target lesions
Units Other Than Participants: lesions
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 151
Number analyzed (lesions) | 201
percentage of target lesions | 0.5 [0.0 to 2.7]

78. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: This measure indicates the absolute change between two timepoints represented by the mean.
  SF-12® Health Survey is validated measure using 12 questions to measure functional health and well-being from the patient's point of view. Scores on the scale are 0% (indicating poor perceived health status) to 100% (indicating excellent perceived health status) possible.
Time Frame: Baseline and 1 month
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 132
score on a scale | 10.4 (11.3)

79. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: as for outcome 78
Time Frame: Baseline and 9 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 136
score on a scale | 9.8 (11.5)

80. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: as for outcome 78
Time Frame: Baseline and 2 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 112
score on a scale | 8.2 (12.7)

81. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: as for outcome 78
Time Frame: Baseline and 3 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 108
score on a scale | 8.9 (13.7)

82. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 78
Time Frame: Baseline and 1 month
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 132
score on a scale | 2.3 (10.7)

83. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 78
Time Frame: Baseline and 9 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 136
score on a scale | 0.9 (11.7)

84. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 78
Time Frame: Baseline and 2 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 112
score on a scale | 2.2 (12.1)

85. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 78
Time Frame: Baseline and 3 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Number analyzed (Participants) | 108
score on a scale | -0.5 (13.4)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Designations were chosen to match Abbott Categories coding and may differ from other coding systems. Denominators for event rates excludes: lost to follow-up, withdrew through 3 years without adverse events (AE). Entries in the AE category column were coded using trial specific in-house coding classification.
Arm/Group | Omnilink Elite™ Peripheral Balloon-Expandable Stent System
Serious Adverse Events (participants affected / at risk) | 94/153
Other Adverse Events (participants affected / at risk) | 84/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omnilink Elite™ Peripheral Balloon-Expandable Stent System (N=153)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) — Access Site Complication per Abbott Vascular (AV) Organ Systems
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) — Access Site Complication per Abbott Vascular (AV) Organ Systems
Anemia (Blood and lymphatic system disorders) | 9 (10)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (11)
Angina (Cardiac disorders) | 2 (2)
Arrhythmias (other than bradycardia) (Cardiac disorders) | 7 (8)
Cardiac / Hemodynamic (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 5 (5)
Myocardial Infarction - Non-Q- wave (Cardiac disorders) | 1 (1)
Myocardial Infarction - Q- wave (Cardiac disorders) | 1 (1)
Other: Arrhythmia (Cardiac disorders) | 1 (1)
Other: Chest Pain (Cardiac disorders) | 1 (1)
Other: Coronary Artery Disease (Cardiac disorders) | 11 (11)
Pain (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) — Cardiac/Hemodynamic
Congestive Heart Failure (Cardiac disorders) | 2 (2) — Cardiac/Hemodynamic
Hypertension (Cardiac disorders) | 3 (6) — Cardiac/Hemodynamic
Hypotension (Cardiac disorders) | 4 (4) — Cardiac/Hemodynamic
Pulmonary Edema (Cardiac disorders) | 1 (1) — Cardiac/Hemodynamic
Syncope (Cardiac disorders) | 3 (3) — Cardiac/Hemodynamic
Diarrhea (Gastrointestinal disorders) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 7 (7)
Gastro-intestinal (Gastrointestinal disorders) | 4 (5)
Infection (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Other: Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Other: Cholecystitis (Gastrointestinal disorders) | 3 (3)
Other: Cholelithiasis (Gastrointestinal disorders) | 1 (1)
Other: Dehydration (Gastrointestinal disorders) | 1 (1)
Other: Diabetic Gastroparesis (Gastrointestinal disorders) | 1 (1)
Other: Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Other: Incisional Hernia (Gastrointestinal disorders) | 1 (1)
Other: Pancreatitis (Gastrointestinal disorders) | 1 (2)
Pain (Gastrointestinal disorders) | 2 (2)
Surgery/Interventional Procedure (Gastrointestinal disorders) | 1 (1)
Gastro-intestinal (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Other: Abscess (Infections and infestations) | 1 (2)
Other: Bronchitis (Infections and infestations) | 1 (1)
Other: Cellulitis (Infections and infestations) | 3 (4)
Pneumonia (Infections and infestations) | 14 (21)
Respiratory (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Wound complication or wound infection (Infections and infestations) | 2 (2)
Other: Acidosis (Metabolism and nutrition disorders) | 1 (1)
Other: Fatigue (Metabolism and nutrition disorders) | 1 (1)
Other: Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Other: Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Other: Hyponatremia (Metabolism and nutrition disorders) | 2 (5)
Edema (non pulmonary) (General disorders) | 2 (2)
Genito-urinary (General disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 16 (17)
Other (General disorders) | 1 (1)
Other: Acquired Spondylolistheses (General disorders) | 1 (1)
Other: Frequent Falls (General disorders) | 1 (1)
Other: Lethargy (General disorders) | 1 (1)
Other: Multi Organ Failure (General disorders) | 1 (1)
Other: Shingles (General disorders) | 1 (1)
Other: Trauma (General disorders) | 1 (1)
Surgery/Interventional Procedure (General disorders) | 1 (1)
Myocardial Infarction - Non-Q- wave (Cardiac disorders) | 2 (2)
Myocardial Infarction - Unknown (Cardiac disorders) | 3 (3)
Other: Myocardial Infarction - Non-Q Wave (Cardiac disorders) | 1 (1)
Mental Status Change (Nervous system disorders) | 3 (4) — Neurologic other than stroke
Other: Anoxic Injury (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Seizure (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Transient Ischemic Attack (Nervous system disorders) | 4 (4) — Neurologic other than stroke
Vision disturbance (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Bleeding (Injury, poisoning and procedural complications) | 1 (1) — Non-Access Site Bleeding
Hematoma (Injury, poisoning and procedural complications) | 1 (1) — Non-Access Site Bleeding
Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1)
Dissection (Injury, poisoning and procedural complications) | 2 (2) — Procedure-related
Distal Emboli (Injury, poisoning and procedural complications) | 1 (1) — Procedure-related
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Other: Acute Exacerbation Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Viral, bacterial and fungal infections (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: CVA (Vascular disorders) | 1 (1) — Stroke
Other: Cerebral Vascular Accident (Vascular disorders) | 2 (2) — Stroke
Other: Lacunar Stroke (Vascular disorders) | 1 (1)
Other: Stroke (Vascular disorders) | 1 (1)
Dissection (Vascular disorders) | 2 (2)
Gastro-intestinal (Vascular disorders) | 1 (1)
Ischemia (Vascular disorders) | 2 (4)
Occlusion (Vascular disorders) | 5 (7)
Other: Aortic Iliac (Vascular disorders) | 1 (1)
Other: Carotid Artery Disease (Vascular disorders) | 1 (1)
Other: Deep Vein Thrombosis (Vascular disorders) | 3 (3)
Other: Peripheral Vascular Disease (Vascular disorders) | 10 (12)
Other: Stenosis (Vascular disorders) | 1 (1)
Pain (Vascular disorders) | 1 (2)
Pulmonary Embolism (Vascular disorders) | 1 (1)
Renal (Vascular disorders) | 1 (1)
Restenosis (Vascular disorders) | 14 (16)
Stenosis (Vascular disorders) | 25 (44)
Stent Thrombosis (Vascular disorders) | 1 (1)
Surgery/Interventional Procedure (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omnilink Elite™ Peripheral Balloon-Expandable Stent System (N=153)
Anemia (Blood and lymphatic system disorders) | 8 (9)
Hypertension (Cardiac disorders) | 8 (9) — Cardiac/Hemodynamic
Edema (non pulmonary) (General disorders) | 13 (15)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 48 (78)
Other: Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Other: Peripheral Vascular Disease (Vascular disorders) | 21 (23)
Stenosis (Vascular disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less